CLINICAL TRIAL: NCT01901029
Title: Prevalence of Reproductive Health Problems and Their Social, Psychological and Physical Association Among Men in Floating Population: a Large-Scale Cross-Sectional Study in Dongguan City
Brief Title: Male Reproductive Health of Floating Population: a Large-Scale Survey in Dongguan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Dongguan Taiping People's Hospital (Unknown)
Responsible Party: Principal Investigator, Wan Zi, Medical Doctor, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: DGFPmrhs
Record Dates: First submitted 2013-07-07; First posted 2013-07-17 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Sexual Behavior; Erectile Dysfunction; Premature Ejaculation
Keywords: Male Reproductive Health; Floating Population; Sexual Behavior; Erectile Dysfunction; Premature Ejaculation
MeSH Terms: conditions — Sexual Behavior; Erectile Dysfunction; Premature Ejaculation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- men of floating population: males who live in Dongguan more than 6 months and without residence cards
- men of non-floating population: males who live in Dongguan more than 6 months and with residence cards

SUMMARY:
To determine the prevalence of sexual problems particularly premature ejaculation and erectile dysfunction among men working in factories of Dongguan city, using the self-rating scales like International Index of Erectile Function, and to investigate the characteristics or risk factors associated with these sexual problems in floating population through regression analysis.

DETAILED DESCRIPTION:
In China, the floating population is a special group of people who work and live outside their hometowns and without residence cards of that area they reside. Sexual problems are common in floating population, majority of whom are in their sex active age. There is a lack of studies concerning these sexual problems, so we conduct this survey to investigate the sexual dysfunctions among men, especially the floating population, and to find out whether most of these sexual problems are related to their social lives, medical illnesses, and psychological status.

ELIGIBILITY:
Inclusion Criteria:

* have reached 18 years old
* live in Dongguan more than 6 months
* floating population
* with or without residence card

Exclusion Criteria:

* younger than 18 years old
* live in Dongguan less than 6 months

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: male workers in several towns of Dongguan city
Sampling Method: Probability Sample
Enrollment: 3100 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of sexual problems | one month
  Determine the prevalence of sexual problems among men of floating population in Dongguan.

SECONDARY OUTCOMES:
Association between risk factors and sexual problems | one month
  Association between social, psychological and physical factors and sexual problems.

CONTACTS AND LOCATIONS:
Overall Officials: Jianbo Ruan, MM, Study Director — Dongguan Taiping People's Hospital
Locations (1):
- Dongguan Taiping People's Hospital Andrology Department, Dongguan, Guangdong, China